CLINICAL TRIAL: NCT02177955
Title: Comparative Study of Hemodynamic Changes Caused by Diazepam and Midazolam During Third Molar Surgery. A Prospective Randomized Study
Brief Title: Comparative Study of Hemodynamic Changes Caused by Diazepam and Midazolam During Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jimmy Barbalho (Other)
Collaborators: University of Pernambuco (Other)
Responsible Party: Sponsor-Investigator, Jimmy Barbalho, DDs, University of Pernambuco
Organization: University of Pernambuco (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 001.0.097.000-08; 001.0.097.000-08 (Other: 001.0.097.000-08)
Record Dates: First submitted 2014-06-21; First posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Anxiety
Keywords: Third Molar; Anty-anxiety drugs; hemodynamic; Benzodiazepines
MeSH Terms: conditions — Anxiety Disorders | interventions — Midazolam; Diazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- midazolan (Placebo Comparator): 7.5 mg midazolan 45 minutes before the surgery
  Interventions: Drug: 7.5 mg Midazolam
- diazepam (Placebo Comparator): 10 mg diazepam 45 minutes before the surgery
  Interventions: Drug: 10 mg diazepam

INTERVENTIONS:
Drug: 7.5 mg Midazolam — 7.5 mg midazolam 45 minutes before surgery
  Arms: midazolan
Drug: 10 mg diazepam — 10 mg midazolam 45 minutes before surgery
  Arms: diazepam

SUMMARY:
Objective: The aim of the present study was to compare hemodynamic changes using 7.5 mg of midazolam and 10.0 mg of diazepam during the surgical removal of symmetrically positioned third molars.

Study design: A prospective, randomized, double-blind, clinical trial was carried out involving 120 patients divided in three groups: Group 1 (diazepam and placebo), Group 2 (midazolam and placebo) and Group 3 (diazepam and midazolam). Each subject underwent two surgeries on separate occasions under local anesthesia.

DETAILED DESCRIPTION:
Study design A double-blind, randomized, crossover, clinical trial with a split-mouth design was carried out. This study received approval from the Human Research Ethics Committee of the institution at which it was carried out (process number: 001.0.097.000-08) and was conducted in compliance with the Consolidated Standards of Reporting Trials (CONSORT) statement. All patients signed a statement of informed consent agreeing to participate in the study.

Sample size and pilot study The sample size was estimated using the a computational program. Thirty patients were submitted to third molar surgeries in a pilot study to determine the sample size. This step was necessary due to the lack of similar studies in the literature. Calculations were performed with specific programs taking into consideration the variables, a 95% confidence interval, 80% test power and 5% error. At the end of the study, 120 patients were analyzed (40 in each group), totaling 240 surgeries.

Sample selection One hundred twenty eight individuals between 18 and 40 years of age were selected for participation in the present study and submission to maxillary and mandibular third molar extractions bilaterally at the Department of Oral-Maxillofacial Surgery. Each patient was to be submitted to two surgeries. The third molars (maxillary or mandibular) needed to have the same degree of impaction on both sides.

Three groups were formed: Group A received diazepam and placebo, Group B received midazolam and placebo and Group C received midazolam and diazepam. For the purposes of randomization and blinding of the surgeon and researcher in charge of analyzing the results, the groups were renominated Groups 1, 2 and 3. The randomization procedure was carried out by a researcher who was not directly involved in the surgeries or evaluations. Sequentially numbered, sealed, opaque envelopes were used, each containing a combination of substances and the side to be submitted to the first surgery. For each patient, the researcher opened an envelope, informed the main investigator and surgeon of the side to be operated, and administered the substance to the patient. The second surgery was performed on the contralateral side with the administration of the second substance. Blinding was performed to avoid awareness regarding what substance was administered in each surgery. For such, the pills were fabricated with the same outer color and a standardized size at the Pernambuco Pharmaceutical Laboratory (Brazil) and were packaged in recipients with the same color. The recipients were denominated 1, 2 and 3.

Surgical procedures and medications As the patients were classified as healthy, no prophylactic use of antibiotics was performed prior to surgery for the prevention of bacterial endocarditis, as recommended by the American Heart Association. All patients rinsed their mouths with 0.12% chlorhexidine for one minute prior to surgery to reduce the bacterial population in the oral cavity. Moreover, all patients were instructed to take two 4-mg pills of dexamethasone one hour prior to surgery. The use of a corticosteroid in the preoperative period minimizes the occurrence of postoperative swelling and reduces the risk of trismus.13 The substances (diazepam, midazolam and placebo) were administered orally 45 minutes prior to the surgical procedure. As the substances were masked, neither the surgeon nor the patient was aware of what substance was given (double-blind study).

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were classification in Group 1 of the American Society of Anesthesiology (normal healthy patient with no adverse systemic condition or continuous use of medication) and no self-reported reactions or allergies to the drugs employed in the study

Exclusion Criteria:

* The exclusion criteria were refusal to participate after reading the statement of informed consent, self-reported allergy to the drugs employed and failure to return for the second surgery on the contralateral side

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in systolic blood pressure until the end of surgery | baseline, 2 minutes, 7 minutes, 12 minutes, end of surgery.
Changes from baseline in diastolic blood pressure until the end of surgery | Baseline, 2 minutes, 7 minutes, 12 minutes, end of surgery
Changes from baseline in mean blood pressure until the end of surgery | Baseline, 2 minutes, 7 minutes, 12 minutes, end of surgery
Changes from baseline in heart rate until the end of surgery | Baseline, 2 minutes, 7 minutes, 12 minutes, end of surgery
Changes from baseline in rate pressure product until the end of surgery | Baseline, 2 minutes, 7 minutes, 12 minutes, end of surgery
  The rate pressure is the product of the multiplication of systolic blood pressure by heart rate
Changes from baseline in oxygen saturation until the end of surgery | Baseline, 2 minutes, 7 minutes, 12 minutes, end of surgery
Change from baseline in pressure rate quotient until the end of surgery | Baseline, 2 minutes, 7 minutes, 12 minutes, end of surgery
  Pressure rate quotient is calculated by dividing mean blood pressure by heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Hécio H De Morais, PhD, Principal Investigator — University of Pernambuco
Locations (1):
- School of Dentistry of Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- See also: Related Info — http://www.upe.br/portal/